CLINICAL TRIAL: NCT06925581
Title: A Phase I/II Clinical Trial to Evaluate the Pharmacokinetics, Radiation Dosimetry, Safety and Preliminary Efficacy of HRS-6768 in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Trial of HRS-6768 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6768-101
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-6768 (Experimental)
  Interventions: Drug: HRS-6768

INTERVENTIONS:
Drug: HRS-6768 — HRS-6768

SUMMARY:
The study is being conducted to evaluate the pharmacokinetics, radiation dosimetry, safety and preliminary efficacy of HRS-6768. To explore the reasonable dosage of HRS-6768 in the treatment of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. subjects with solid tumors who have been histologically or cytologically diagnosed with advanced - stage (unresectable or metastatic) disease, have failed standard treatment (disease progression or intolerance), or lack effective treatment methods.
3. There must be at least one evaluable lesion .
4. ECOG 0-1
5. The functions of major organs are in good condition.

Exclusion Criteria:

1. The patient has experienced significant weight loss within 28 days prior to signing the informed consent form.
2. The patient has previously received radiopharmaceutical therapy or radioactive embolization, or has previously undergone any external beam radiotherapy (EBRT) involving more than 25% of the bone marrow, or has previously had EBRT directly applied to the kidneys, or has received any EBRT within 2 weeks before the first dose.
3. The patient has received anti - tumor treatments such as surgery (excluding diagnostic biopsy and serous cavity effusion drainage), checkpoint inhibitor therapy, other antibody therapies, chemotherapy, targeted therapy, gene therapy, and vaccine therapy within 4 weeks before the first dose.
4. The patient has had a severe infection (CTCAE > Grade 2) within 4 weeks before the first dose, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications. The patient has had symptoms and signs of infection within 2 weeks before the first dose that require intravenous antibiotic treatment (excluding cases of prophylactic antibiotic use).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1:Dose-limiting toxicity (DLTs) | From first dose of study drug through at least 6 weeks
  To evaluate the safety and tolerability of HRS-6768 and determine the RP2D.
Phase 1: recommended Phase 2 dose (RP2D) | From first dose of study drug to end of phase 1 treatment (up to approximately 1 years)
  To evaluate the safety and tolerability of HRS-6768 and determine the RP2D.
Phase 1: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of HRS-6768 | From first dose of study drug to end of treatment (up to approximately 2 years)
  Phase 1: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of HRS-6768
Phase 2: Progression-free survival (PFS) | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)

SECONDARY OUTCOMES:
Phase 1/2: Absorbed dose (Gy) estimated in organs and tumor lesions | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  To measure the radiation dosimetry of HRS-6768
Phase 1/2: Cmax of HRS-6768 | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  To evaluate the PK of HRS-6768
Phase 1/2: Tmax of HRS-6768 | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  To evaluate the PK of HRS-6768
Phase 1/2: Area under the curve (AUC) of HRS-6768 | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  To evaluate the PK of HRS-6768
Phase 1/2: clearance (CL) of HRS-6768 | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  To evaluate the PK of HRS-6768
Phase 1/2: Objective Response Rate (ORR) | From first dose of study drug until disease progression or end of treatment (up to approximately 1 years)
  Objective response is defined as a best confirmed response of CR or PR by RECIST v1.1 as assessed by the investigator.
Phase 1/2: Duration of Response (DoR) | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
Phase 1/2: Disease Control Rate (DCR) | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  Disease Control Rate (DCR) is defined as the frequency and percentage of participants with stable disease (SD) or CR or PR.
Phase 1: Progression-free survival (PFS) | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  Progression-free survival (PFS) is defined as the time from the date of first dose to the date of first evidence of radiographic progression or death due to any cause, whichever occurred first.
Phase 1/2: Overall Survival (OS) | From first dose of study drug until disease progression or end of treatment (up to approximately 2 years)
  Overall Survival (OS) is defined as the time from the date of first dose to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gaobo Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided